CLINICAL TRIAL: NCT04422470
Title: Observational Prospective Cohort Study - Registry of Patients With Hematologic Disease and COVID-19 in Russia (CHRONOS19)
Brief Title: Registry of Patients With Hematologic Disease and COVID-19 in Russia
Acronym: CHRONOS19
Status: Completed | Type: Observational
Sponsor: National Research Center for Hematology, Russia (Network)
Collaborators: Foundation for Cancer Research Support (RakFond) (Unknown); Enrollme.ru, LLC (Network)
Responsible Party: Sponsor
Other Study IDs: CHRONOS19
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus Infection and Hematologic Diseases
Keywords: COVID-19; Blood diseases; Leukemia; Lymphoma
MeSH Terms: conditions — Coronavirus Infections; Hematologic Diseases; COVID-19; Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional study — Non-interventional study

SUMMARY:
This is an observational prospective cohort study to evaluate the clinical course and outcomes of COVID-19 and the underlying disease in patients with hematologic disease (malignant or non-malignant).

DETAILED DESCRIPTION:
This is a web-based registry. After registration, physicians from hematology clinical centers and hospitals in Russia will receive access to the web platform for clinical trial management to fill in the online data collection form in a de-identified manner. This form includes questions about general clinical history of hematologic disease, manifestation, treatment, and the course of COVID-19, concomitant conditions, consequences on the hematologic disease, short-term and long-term outcomes. It will take approximately 10 min to answer the questions. Patients will be followed for 30 days after COVID-19 diagnosis and up to 6 months for hematologic disease outcomes and overall survival assessment.

ELIGIBILITY:
Inclusion Criteria

* Age 18 or older
* Any previously or currently diagnosed hematologic disease
* Laboratory confirmed or suspected (based on clinical symptoms and/or CT) COVID-19
* Known outcome of COVID-19 in case of retrospective data input (protocol allows retrospective data input for patients who were prospectively followed in local centers)

Exclusion Criteria

• Loss of follow-up within 30 days after COVID-19 diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hematologic disease (both malignant and non-malignant) infected with SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 666 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
30-day all-cause mortality | 30 day
  Rate of death from any cause

SECONDARY OUTCOMES:
COVID-19 complications | 30 day
  Rate of COVID-19 complications
ICU admission | 30 day
  Rate of ICU admission
Mechanical ventilation / O2 requirement | 30 day
  Rate of mechanical ventilation / O2 requirement
Relapse or progression of hematologic disease | 30 day, 90 day and 180 day
  Rate of relapse or progression of hematologic disease
Overall survival | 30 day, 90 day and 180 day
  Number of patients alive
Risk factors | 30 day, 90 day and 180 day
  Putative risk factors for the severity and lethality of COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Elena Parovichnikova, Study Chair — National Research Center for Hematology
Locations (15):
- Russia (15):
  - Republican Clinical Hospital of Tatarstan, Kazan'
  - City Hospital n.a. V.V. Veresaev, Moscow
  - Clinical Hospital n.a. S.P. Botkin, Moscow
  - N.V. Sklifosovsky Emergency Institute, Moscow
  - National Research Center for Hematology, Moscow
  - Regional Clinical Hospital N.A. Semashko, Nizhny Novgorod
  - Regional Hospital, Novosibirsk
  - Regional Clinical Hospital, Omsk
  - RM Gorbacheva Research Institute of Pediatric Oncology, Hematology and Transplantation, Pavlov University, Saint Petersburg
  - Republican Clinical Hospital No4, Saransk
  - Republic Clinical Hospital n.a. N.A. Semashko, Ulan-Ude
  - Regional Clinical Hospital, Vladimir
  - Regional Clinical Hospital No2, Vladivostok
  - Regional Clinical Hospital, Yaroslavl
  - Regional Clinical Hospital No1, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No